CLINICAL TRIAL: NCT02960464
Title: Transcranial Direct Current Stimulation for Treatment of Depression in Parkinson's Disease, a Randomized Placebo-controlled Clinical Trial
Brief Title: tDCS for Treatment of Depression in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Santa Marcelina (Other)
Responsible Party: Principal Investigator, Pedro Caldana Gordon, Principal Investigator, Hospital Santa Marcelina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSMarcelina
Record Dates: First submitted 2016-11-08; First posted 2016-11-09 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Idiopathic Parkinson Disease; Depression
Keywords: Parkinson Disease; Depression; Transcranial Direct Current Stimulation; Neuromodulation
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Arm (Active Comparator): Active sessions will involve the placement of the anode over the scalp corresponding to the F3 (10-20 EEG system), and cathode over F4. Current intensity will be 2mA, and the stimulation will last for 20 minutes.
  Interventions: Device: Transcranial direct current stimulation
- Sham Arm (Sham Comparator): Sham stimulation will follow the same procedure as the Active, however after 30 seconds of stimulation, the current is turned off, mimicking the initial sensation of the tDCS session but providing no clinical or physiological effect.
  Interventions: Device: Sham Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation
  Arms: Active Arm
Device: Sham Transcranial direct current stimulation
  Arms: Sham Arm

SUMMARY:
Investigation of possible benefits of transcranial direct current stimulation (tDCS) as a treatment of depression in patients with Parkinson's Disease, through a randomized placebo-controlled clinical trial.

DETAILED DESCRIPTION:
We aim to investigate the effects of transcranial direct current stimulation (tDCS) as treatment for depression in patients with Parkinson's Disease. We have designed a clinical trial in which volunteers that fulfill inclusion criteria will receive 15 sessions of tDCS during 1 week (3 sessions a day, with 30 minutes interval in between). Subjects will be randomly allocated into two groups, one that will receive the real intervention (active) and the other that will receive the placebo intervention (sham). The collaborator in charge of administering the session will not participate in the evaluations, keeping both subjects and evaluators blinded to the nature of the sessions. Subjects will be evaluated at baseline, and after the end of sessions, 1 week, 4 weeks and 8 weeks, the latter being the main outcome.

We aim to enroll 50 subjects, 25 for each arm. The sample size calculation took into consideration previous clinical trials using tDCS for depression in different settings.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease
* Geriatric Depression Scale - 15 higher that 5
* Major Depression Disorder

Exclusion Criteria:

* CNS disease other than Parkinson's Disease (i.e. epilepsy, stroke)
* Mental disorder other than depression on anxiety disorder (i.e. bipolar disorder, schizophrenia)
* Previous neurosurgical intervention (i.e. DBS)
* Current use of antidepressant drug
* High suicidality risk
* Limited capacity of understanding written and spoken Portuguese

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | 8 weeks

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale | 8 weeks
Mini-Mental State Examination | 8 weeks
Hamilton Anxiety Rating Scale | 8 weeks
Geriatric Depression Scale -15 | 8 weeks
Parkinson's Disease Questionnaire - 39 | 8 weeks
Lille apathy rating scale | 8 weeks
Quantitative EEG | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Sheila Rocha, MD, PhD, Study Director — Hospital Santa Marcelina
Locations (1):
- Hospital Santa Marcelina, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No